CLINICAL TRIAL: NCT02653664
Title: Hypnosis and Meditation for Pain Management in Veterans: Efficacy and Mechanisms
Brief Title: Chronic Pain Skills Study
Acronym: CPSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency); Washington State University (Other)
Responsible Party: Principal Investigator, Mark Jensen, Professor, Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 49799
Record Dates: First submitted 2015-12-10; First posted 2016-01-12 (Estimated); Results first posted 2021-10-18 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Sleep
MeSH Terms: conditions — Chronic Pain | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Condition #1: PsychoEducation (ED) (Experimental): Condition #1 will include 8 90-minute group sessions that will educate the subject about chronic pain, discuss the impact of pain, and inform the subject of different ways to manage it in hopes of decreasing pain and its impact on the subject's life. Participants in this condition will be given pre-recorded audio recordings of the content of the sessions to listen to.
  Interventions: Behavioral: PsychoEducation
- Condition #2:Self-Hypnosis Training (HYP) (Experimental): In condition #2, the facilitator will perform a standard hypnotic short induction followed by therapeutic suggestions, including post-hypnotic suggestions. Participants will relax in a comfortable position with their eyes closed and will simply listen to the clinician read a standardized hypnotic script that will include an induction followed by suggestions for decreased pain and improvement in co-morbid symptoms (e.g., improved mood and optimism, relaxation, sleep quality).
  Interventions: Behavioral: Self-Hypnosis Training
- Condition #3: Mindfulness Meditation (MM) (Experimental): In condition #3, the facilitator will teach participants Vipassana meditation, which is the specific form of mindfulness meditation (MM) typically implemented in mindfulness research. The emphasis is placed upon developing focused attention on an object of awareness, such as the breath. This focus is then expanded to include a more open, non-judgmental monitoring of any sensory, emotional, or cognitive events. Time will also be devoted to problem solving around any difficulties with MM practice.
  Interventions: Behavioral: Mindfulness Meditation

INTERVENTIONS:
Behavioral: PsychoEducation — Condition #1
  Arms: Condition #1: PsychoEducation (ED)
Behavioral: Self-Hypnosis Training — Condition #2
  Arms: Condition #2:Self-Hypnosis Training (HYP)
Behavioral: Mindfulness Meditation — Condition #3
  Arms: Condition #3: Mindfulness Meditation (MM)

SUMMARY:
Chronic pain is a significant problem for many Veterans, including new Veterans returning from Iraq and Afghanistan. It is also associated with a number of other significant problems, such as post-traumatic stress disorder and sleep problems. All of these can have significant negative effects of the quality of life of Veterans

Three different types of treatment that have been used to treat chronic pain in the general population include self-hypnosis, education about chronic pain, and teaching individuals how to be more mindful. The purpose of this study is to see if these three treatments can help decrease pain in Veterans. Additionally, the researchers want to determine if each of these treatments can help reduce the negative consequences associated with pain, such as changes in mood, sleep, and enjoyment of life.

Different types of treatment that include self-hypnosis, education about chronic pain, and learning skills on how to change how a person perceives his/her pain have been used to treat chronic pain the general population.

The purpose of this study of this study is to see if these different treatments can help decrease pain and improve quality of life in Veterans with chronic pain, and determine how and why these treatments are effective. A subject must have a Veteran status, have chronic pain, speak English and be at least 18 years old to participate.

Sleep Sub-Study

Chronic pain and sleep problems are common among Veterans. Study researchers believe the treatment interventions provided as part of the main study will help improve pain and sleep. However, the main study does not include a "real time" measurement of sleep nor does it include any specific strategies for examining the relationship between sleep and pain.

Previous research has shown that adequate sleep has been linked to improvements in pain reports. Adversely, sleep deprivation has been found to increase pain perception since it decreases a person's ability to disengage from pain. Therefore, the purpose of this sub-study is to measure sleep in order to learn more about how it interacts with chronic pain.

All of the subjects in this sub-study will be Veterans recruited from VA Puget Sound who experience moderate-to-severe chronic pain on a regular basis and who have enrolled in the main study. Study investigators will enroll up to 135 subjects into the sub-study.

DETAILED DESCRIPTION:
Cognitive Assessment

Following enrollment, research staff will administer a battery of five neuropsychological measures assessing memory, information processing, and executive functioning. These measures take approximately 20-30 minutes to complete.

Hypnotic and Relaxation Exercise

A research staff member will administer in person the Modified Stanford Hypnotic Clinical Scale (SHCS) to assess hypnotizability for all participants following enrollment but prior to randomization. This measure takes approximately 15-20 minutes to complete.

Baseline Data and Demographic Form

A research staff member will then ask the participant to provide demographic data (age, sex, marital status, income, education level, employment status) and deployment history (number and month of deployments, whether deployment involved hostile duty) for descriptive purposes. Study investigators will also ask participants their history of receiving the study treatments, and the presence of history of military sexual trauma.

The baseline data and demographic form will take approximately 20-30 minutes to complete, and may be completed following enrollment either in person or over the telephone at a later time if more convenient for the participant.

Brain Wave Activity (or EEG) Assessment

Brain wave activity will be assessed following enrollment by conducting a brain wave activity or EEG assessment. The brain wave activity assessment will take place at the Integrated Brain Imaging Center (IBIC) at the University of Washington main campus. The IBIC is a research-dedicated technology center organized under the department of Radiology.

EEG will be sampled with an electrode array using an electrode net dipped in a saline solution. The research staff member, an IBIC employee with a Without Compensation (WOC) appointment at the VA Puget Sound Health Care System (VAPSHCS), will collect the EEG activity data, and ask the participant to remain as still as possible during portions of the assessment.

The EEG technician will collect from the participant data regarding medication used within 24 hours of assessment. He/she will also ask the participant to rate the intensity of his or her pain just before the assessment (current pain), after a few minutes of the assessment (current pain and worst, least, and average pain over the past few minutes), and at the end of the EEG session (current pain, and worst, least, and average pain over the past few minutes), using 0-10 Numerical Rating Scales.

The entire brain wave activity assessment will take approximately 45-60 minutes to complete. Subjects will be asked to complete the same brain activity assessment following completion of treatment following the same procedures above. Participants may still participate in the study if they decline to participate in the EEG assessments.

Assessment: Pre-Treatment and General Overview

Subjective reports of pain intensity vary over time, and to most accurately measure pain intensity (our primary outcome), it is most valid to assess multiple times and take an average. Hence, study investigators have developed a method of assessment that will seek to obtain up to four telephone assessments over a period of one week or 7 days with a minimum of 24 hours between each assessment. During each telephone contact, research staff will ask participants, at minimum, to rate their current, average, worst and least pain intensity over the past 24 hours, as well as their average pain intensity over the past 7 days. In addition, if possible, research staff will ask the participant to rate their current, average, worst and least pain intensity over the past week during the final telephone contact. These assessments will be referred to as "short assessments." The primary outcome will be an average of all of the 24-hour ratings (range=1-4 ratings) of average pain intensity obtained over a period of one week during each assessment period.

In addition, sometime during this assessment period researchers will ask questions regarding pain interference, depression, anxiety, sleep disturbance, post-traumatic stress disorder (PTSD) symptoms, medication use, medical services utilization, thoughts about pain and treatment motivation. This latter set of questions will only be asked once during the assessment period, and will be referred to as "the long assessment." Research staff will give participants the option to: 1) complete the long assessment during one of the four short telephone assessments described above; or 2) spread the long assessment across several days during the assessment period. The entire long assessment or portions thereof may fall up to two days outside the 7-day period for the four short assessments.

The entire time required to answer questions during the assessment period is 45-60 minutes.

The assessment period described above will be completed prior to initiating treatment, and then after completion of treatment sessions #2, 4 and 6 and 8 (i.e. post-treatment), and 3 and 6 months following the end of treatment for a total of seven times. These assessment periods that occur following the start of treatment will also include questions about group climate, therapeutic alliance with the group clinician, treatment satisfaction, and overall improvement since the participant began the pain program.

Randomization

Enrolled participants who complete the required baseline components (cognitive assessment, hypnotic and relaxation exercise, baseline data form, and pre-treatment assessment period) will be randomized in stratified blocks to ensure that participants with each sex and pain type (neuropathic, non-neuropathic, mixed or undetermined) have an equal chance of being randomized to one of the 3 conditions.

Treatment Scheduling

Cohorts of study intervention groups will be offered beginning every four months. In each 4-month period, there will be two class options for each condition, one based in Seattle and one at American Lake. Thus, there will be six classes offered per four month period, or a total of 18 classes per year.

Up to 15 participants can be enrolled in each intervention class; 10 spots will be protected for research participants, and the remaining 5 for Veterans who have completed the study and wish to try another type of intervention, or who are non-research participants. If any protected research spots are not filled at the start of a cohort, non-research participants will be offered those spots and vice versa.

Treatment

In all three treatment conditions, intervention appointments will be scheduled in regular group clinics at the VA facility (American Lake or Seattle). This means that treatment sessions will appear on the Veterans' lists of regular clinical appointments. Although the appointments are scheduled for 90 minutes, in practice they will last 60-80 minutes, with a 10 minute time cushion built in to allow for participants who may have mobility limitations to arrive, settle, and then vacate the group rooms without hurrying.

The group sessions will be conducted by VAPSHCS providers who have undergone a formal two-day training process that prepares clinicians to conduct each of the three treatment interventions in a group setting.

In all conditions, home practice activities will be assigned to increase engagement in the treatment. Participants will be asked to record the extent of engagement in these activities using a form provided to them by the clinician. Study investigators realize that adherence to interventions assigned outside of treatment sessions may influence study outcomes so will utilize data collected by the clinicians about homework compliance. In addition, all participants in all interventions will be given a treatment workbook with materials to refer to and discuss during the group sessions as well as additional materials to read between sessions.

Please see below for description of study treatment interventions.

Data Collected during Treatment Sessions

Participants will complete and hand in a form regarding their completion of tasks or "homework" assigned by the clinician from the previous session.

In addition, participants will complete and hand in forms before and after each session that include questions regarding pain intensity and comfort level, as well as questions about what the participants have found helpful or non-helpful about the treatment. Finally, study clinicians will complete a form each session that captures information regarding the perceived engagement of each participant in that particular session. All of these forms will be labeled with a subject's name.

Audio Recordings

The group treatment sessions will be audio recorded to make sure the study clinician is following study procedures.

Optional Assessments

For the pre-treatment and post-treatment telephone assessment periods, research staff will use a script to invite participants upon completing the assessment period to participate in an optional assessment consisting of two measures developed by study researchers. The optional assessment should take approximately 10-15 minutes to complete, and consists of questions about how participants feel when they feel pain or think about their pain problem, and how participants respond to their pain.

Open Label Phase

Following the completion of the 6-month telephone assessment period research staff will invite participants to complete in one or both of the treatment groups they did not attend during participation in the main phase. Participants would only participate in one treatment group at a time. The open label phase does not include any screening procedures; all research participants are welcome to participate. Research staff will schedule a consent session if the participant is interested in participating in the 'open label phase' of the study.

Sleep Sub-Study

Subjects enrolled in the main study will be offered the opportunity to participate concurrently in the sleep sub-study. All subjects enrolled in the main study are eligible to participate in the sub-study. Interested subjects will participate in a separate informed consent process before participating in sub-study procedures.

Telephone Assessments

A research staff member will ask each sub-study subject two questions about how much the subject agrees with certain statements about his/her sleep, as well as two questions about how confident the subject is about carrying our certain sleep behaviors. These questions will be asked during the pre-treatment assessment period, 4-week assessment period, post-treatment assessment period, and the assessment period that takes place 3 months following the end of treatment.

Sleep Diary

Three times during his/her participation in the sub-study, study investigators will ask the subject to keep a sleep diary: once following enrollment but prior to randomization, once following the end of treatment, and once three months following the end of treatment. The subject will complete a diary entry twice a day (morning and night) for seven days. In the morning, the subject would answer basic questions about his/her sleep during the previous night, including time the subject thinks s/he fell asleep, the quality of his/her sleep, and any other experiences that might have affected his/her sleep. In the evening, the subject will answer questions about how the subject felt that day, any problems s/he experienced such as illness or discomfort, and basic activities s/he participated in like going to work, napping, drinking caffeinated beverages, etc.

Also, the subject will be instructed to call a toll free number twice a day to report when s/he woke up in the morning, and when s/he is going to sleep in the evening.

Actigraphy Device

Three times during his/her participation in the sub-study, study investigators will ask the subject to wear a sleep monitor device called an Actigraph: once following enrollment but prior to randomization, once following the end of treatment, and once three months following the end of treatment. The subject would wear the actigraph (Actiwatch , Philips Respironics, Bend, OR) like a wrist watch on his/her non-dominant arm. The device will measure how long the subject sleeps, as well as the overall quality of his/her sleep. The subject will wear the actigraph at all times during the same 7-day period s/he is completing the sleep diary except for when the subjects is participating in activities that might get the actigraph wet like swimming, showering, or bathing.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. Veteran eligible for services through Veteran Health Affairs;
3. experience moderate to severe chronic pain on a regular basis; and
4. able to read, speak and understand English.

Exclusion Criteria:

1. severe cognitive impairment;
2. current or history of psychiatric or behavioral issues that require immediate attention and/or prevent the subject from participating effectively in the study;
3. reported use of a high dose of an opioid(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2015-10-09 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jensen, PhD, Principal Investigator — University of Washington; Rhonda Williams, PhD, Principal Investigator — VA Puget Sound Healthcare System (VAPSHCS)
Locations (5):
- United States (5):
  - University of Washington, Ninth and Jefferson Building, Seattle, Washington
  - University of Washington- Harborview Medical Center, Seattle, Washington
  - VA Puget Sound Health Care System, Seattle Division, Seattle, Washington
  - University of Washington, Integrated Brain Imaging Center, Seattle, Washington
  - VA Puget Sound Health Care System, American Lake, Tacoma, Washington

REFERENCES:
- [Derived] Jensen MP, Ciol MA, Gertz KJ, Ehde DM, Hakimian S, Day MA, Pettet MW, Turner AP, Sarabosing CG, Williams RM. Potential mediators of the effects of clinical hypnosis, mindfulness meditation, and pain education on chronic pain in Veterans. J Pain. 2026 Jan 6;41:106176. doi: 10.1016/j.jpain.2025.106176. Online ahead of print. PMID 41506354
- [Derived] Ho EJ, Turner AP, Jensen MP, Day MA, Ehde DM, Anastas TM, Williams RM. Positive impacts of psychological pain treatments: Supplementary analyses of a randomized clinical trial. Rehabil Psychol. 2025 Feb;70(1):36-45. doi: 10.1037/rep0000557. Epub 2024 Mar 28. PMID 38546554
- [Derived] Anastas TM, Turner AP, Ho EJ, Day MA, Ehde DM, Jensen MP, Williams RM. Evaluating the benefits of a second pain treatment following a clinical trial. Rehabil Psychol. 2024 Feb;69(1):74-83. doi: 10.1037/rep0000510. Epub 2023 Jun 19. PMID 37338442
- [Derived] Turner AP, Edwards KA, Jensen MP, Ehde DM, Day MA, Williams RM. Effects of hypnosis, mindfulness meditation, and education for chronic pain on substance use in veterans: A supplementary analysis of a randomized clinical trial. Rehabil Psychol. 2023 Aug;68(3):261-270. doi: 10.1037/rep0000507. Epub 2023 Jun 8. PMID 37289535
- [Derived] Williams RM, Day MA, Ehde DM, Turner AP, Ciol MA, Gertz KJ, Patterson D, Hakimian S, Suri P, Jensen MP. Effects of hypnosis vs mindfulness meditation vs education on chronic pain intensity and secondary outcomes in veterans: a randomized clinical trial. Pain. 2022 Oct 1;163(10):1905-1918. doi: 10.1097/j.pain.0000000000002586. Epub 2022 Jan 25. PMID 35082248
- [Derived] Turner AP, Jensen MP, Day MA, Williams RM. Behavioral activation and behavioral inhibition: An examination of function in chronic pain. Rehabil Psychol. 2021 Feb;66(1):57-64. doi: 10.1037/rep0000316. Epub 2020 Mar 9. PMID 32150432
- [Derived] Williams RM, Ehde DM, Day M, Turner AP, Hakimian S, Gertz K, Ciol M, McCall A, Kincaid C, Pettet MW, Patterson D, Suri P, Jensen MP. The chronic pain skills study: Protocol for a randomized controlled trial comparing hypnosis, mindfulness meditation and pain education in Veterans. Contemp Clin Trials. 2020 Mar;90:105935. doi: 10.1016/j.cct.2020.105935. Epub 2020 Jan 9. PMID 31926321

RESULTS

PARTICIPANT FLOW:
Period: Post-Treatment
Arm/Group | Condition #1: PsychoEducation (ED) | Condition #2:Self-Hypnosis Training (HYP) | Condition #3: Mindfulness Meditation (MM)
Started (Fifteen of the 343 enrolled subjects withdrew or were withdrawn from the trial prior to randomization. As a result, 328 of the 343 enrolled subjects were randomized. All randomized subjects were listed as 'started' for all time periods following randomization given we conducted an Intention-to-Treat (ITT) analysis.) | 110 | 110 | 108
Primary and Secondary Data | 93 | 104 | 91
Primary Outcome Data Only | 3 | 0 | 3
Completed (Number of subjects who provided average pain intensity data during this assessment period.) | 96 | 104 | 94
Not Completed | 14 | 6 | 14
Not completed — Withdrawal by Subject | 6 | 5 | 7
Not completed — Lost to Follow-up | 8 | 1 | 7
Period: 3 Month Follow-Up
Arm/Group | Condition #1: PsychoEducation (ED) | Condition #2:Self-Hypnosis Training (HYP) | Condition #3: Mindfulness Meditation (MM)
Started (All randomized subjects were listed as 'started' for all time periods following randomization given we conducted an Intention-to-Treat (ITT) analysis.) | 110 | 110 | 108
Primary and Secondary Data | 83 | 95 | 82
Primary Outcome Data Only | 6 | 0 | 1
Completed (Number of subjects who provided average pain intensity data during this assessment period.) | 89 | 95 | 83
Not Completed | 21 | 15 | 25
Not completed — Withdrawal by Subject | 9 | 5 | 9
Not completed — Lost to Follow-up | 9 | 8 | 16
Not completed — Investigator Withdrawn, Behavioral Issues | 0 | 2 | 0
Not completed — Subject Declined Assessment Period, Remained Enrolled in Trial | 3 | 0 | 0
Period: 6 Month Follow-Up
Arm/Group | Condition #1: PsychoEducation (ED) | Condition #2:Self-Hypnosis Training (HYP) | Condition #3: Mindfulness Meditation (MM)
Started (All randomized subjects were listed as 'started' for all time periods following randomization given we conducted an Intention-to-Treat (ITT) analysis.) | 110 | 110 | 108
Primary and Secondary Outcome Data | 85 | 87 | 83
Primary Outcome Data Only | 2 | 2 | 2
Completed (Number of subjects who provided average pain intensity data during this assessment period.) | 87 | 89 | 85
Not Completed | 23 | 21 | 23
Not completed — Withdrawal by Subject | 13 | 7 | 14
Not completed — Lost to Follow-up | 10 | 11 | 9
Not completed — Investigator Withdrawn, Behavioral Issues | 0 | 2 | 0
Not completed — Subject Declined Assessment Period | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Condition #1: PsychoEducation: Condition #1 will include 8 90-minute group sessions that will educate the subject about chronic pain, discuss the impact of pain, and inform the subject of different ways to manage it in hopes of decreasing pain and its impact on the subject's life. Participants in this condition will be given pre-recorded audio recordings of the content of the sessions to listen to.
  PsychoEducation: Condition #1
- Condition #2:Self-Hypnosis Training: In condition #2, the facilitator will perform a standard hypnotic short induction followed by therapeutic suggestions, including post-hypnotic suggestions. Participants will relax in a comfortable position with their eyes closed and will simply listen to the clinician read a standardized hypnotic script that will include an induction followed by suggestions for decreased pain and improvement in co-morbid symptoms (e.g., improved mood and optimism, relaxation, sleep quality).
  Self-Hypnosis Training: Condition #2
- Condition #3: Mindfulness Meditation: In condition #3, the facilitator will teach participants Vipassana meditation, which is the specific form of mindfulness meditation (MM) typically implemented in mindfulness research. The emphasis is placed upon developing focused attention on an object of awareness, such as the breath. This focus is then expanded to include a more open, non-judgmental monitoring of any sensory, emotional, or cognitive events. Time will also be devoted to problem solving around any difficulties with MM practice.
  Mindfulness Meditation: Condition #3
- Total: Total of all reporting groups
Arm/Group | Condition #1: PsychoEducation | Condition #2:Self-Hypnosis Training | Condition #3: Mindfulness Meditation | Total
Number analyzed (Participants) | 110 | 110 | 108 | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (13.5) | 51.0 (12.6) | 55.0 (13.0) | 53.2 (13.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender, n: Men | 80 | 81 | 80 | 241
  Gender, n: Women | 27 | 29 | 28 | 84
  Gender, n: Transgender | 3 | 0 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 10 | 14 | 30
  Not Hispanic or Latino | 101 | 97 | 91 | 289
  Unknown or Not Reported | 3 | 3 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 2 | 8
  Asian | 3 | 2 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 19 | 23 | 16 | 58
  White | 68 | 71 | 68 | 207
  More than one race | 11 | 5 | 13 | 29
  Unknown or Not Reported | 5 | 6 | 4 | 15
Education Level [Count of Participants; unit: Participants]
  High School or Less | 11 | 9 | 6 | 26
  Some College/Technical | 48 | 54 | 52 | 154
  College Degree or Higher | 51 | 47 | 50 | 148
Employment Status [Count of Participants; unit: Participants] — Participants can be represented in more than one employment status category.
  Participants
    Unemployed | 54 | 48 | 36 | 138
    Retired | 45 | 42 | 47 | 134
    Employed Full/Part Time | 26 | 32 | 30 | 88
    Student Full/Part Time | 4 | 4 | 9 | 17
    Home Maker | 6 | 7 | 4 | 17
Married, Living with Partner [Count of Participants; unit: Participants] | 67 | 60 | 55 | 182
Homeless in Past Six Months [Count of Participants; unit: Participants] | 3 | 3 | 2 | 8
Type of Pain [Count of Participants; unit: Participants]
  Probable Neuropathic | 58 | 53 | 49 | 160
  Probable Non-Neuropathic | 27 | 26 | 27 | 80
  Uncertain | 25 | 31 | 32 | 88
Very Good/ Excellent Health [Count of Participants; unit: Participants] | 12 | 8 | 12 | 32
Prior Pain Education [Count of Participants; unit: Participants] | 50 | 42 | 36 | 128
Prior Experience in Hypnosis [Count of Participants; unit: Participants] | 17 | 24 | 27 | 68
Prior Experience in Meditation [Count of Participants; unit: Participants] | 64 | 63 | 62 | 189
Average Pain Intensity [Mean (Standard Deviation); unit: scores on a scale] — An average of all of the 24-hour ratings (range=1-4 ratings) of average pain intensity obtained over a period of one week prior to randomization.
  Range: 0-10, 0='no pain' and 10 ='pain as bad as you can imagine'
  scores on a scale | 5.8 (1.6) | 5.7 (1.8) | 5.9 (1.6) | 5.8 (1.7)
Worst Pain Intensity [Mean (Standard Deviation); unit: scores on a scale] — An average of all of the 24-hour ratings (range=1-4 ratings) of worst pain intensity obtained over a period of one week during each assessment period.
  Range: 0-10, 0='no pain' and 10 ='pain as bad as you can imagine'
  scores on a scale | 7.3 (1.6) | 7.0 (1.8) | 7.2 (1.6) | 7.2 (1.7)
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Instrument [Mean (Standard Deviation); unit: T-score] — This instrument measures the self-reported impact of pain on different aspects of a participant's life.
  The T-score rescales the raw sum score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. A higher score represents more pain interference.
  T-score | 64.6 (5.0) | 63.4 (5.0) | 64.0 (5.8) | 64.0 (5.3)
PROMIS Sleep Disturbance Instrument [Mean (Standard Deviation); unit: T-score] — Per PROMIS, this instrument measures "...self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep."
  The T-score rescales the raw sum score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. A higher score represents more sleep disturbance.
  T-score | 59.2 (8.5) | 59.0 (8.5) | 57.9 (9) | 58.7 (8.7)
PROMIS Anxiety Instrument [Mean (Standard Deviation); unit: T-score] — Per PROMIS: "The PROMIS Anxiety instruments measure self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness)."
  The T-score rescales the raw sum score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. A higher score represents more anxiety.
  T-score | 58.4 (8.9) | 57.0 (9.5) | 57.2 (9.3) | 57.5 (9.2)
PROMIS Depression Instrument [Mean (Standard Deviation); unit: T-score] — Per PROMIS: "The PROMIS Depression instruments assess self-reported negative mood (sadness, guilt), views of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose)."
  The T-score rescales the raw sum score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. A higher score represents more depression.
  T-score | 55.6 (8.8) | 54.1 (9.3) | 53.4 (8.9) | 54.4 (9.0)
Posttraumatic Stress Disorder Checklist (PCL-5) Score [Mean (Standard Deviation); unit: scores on a scale] — The PCL-5 is a 20-item self-report measure reflecting DSM-IV symptoms of PTSD. A total symptom severity score (range = 0-80) can be obtained by summing the scores from each of the 20 items that have response options ranging from 0 "Not at all" to 4 "Extremely." A higher score denotes more severe symptoms of PTSD.
  scores on a scale | 34.3 (17.4) | 32.6 (18.6) | 31.4 (17.3) | 32.8 (17.8)
Classified As Having PTSD [Count of Participants; unit: Participants] | 63 | 53 | 49 | 165
Any Opioid Analgesic Use, Baseline [Count of Participants; unit: Participants] | 35 | 19 | 30 | 84
Morphine Equivalent Dose [Mean (Standard Deviation); unit: milligrams, morphine equivalent] | 6.0 (15.3) | 5.9 (20.6) | 6.3 (16.1) | 6.2 (17.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-Treatment in Average Pain Intensity on a 0-10 Numerical Rating Scale Immediately Following End of Treatment (Post-Treatment)
Description: An average of all of the 24-hour ratings (range=1-4 ratings) of average pain intensity was obtained over a period of one week during each assessment period, pre-treatment and post-treatment.
  Range: 0-10, 0='no pain' and 10 ='pain as bad as you can imagine'
  The difference between the two average scores from the different assessment periods (pre-treatment and post-treatment) was computed by subtracting the pre-treatment score from the post-treatment score, resulting in a change score. A negative value denotes a decrease in pain intensity between the two assessment periods, whereas a positive value denotes an increase.
Time Frame: Change in Average Pain Intensity from Pre-Treatment to Immediately Following End of Approximately Eight Weeks of Treatment (Post-Treatment)
Population: Intent to treat population (all participants assigned to one of the three interventions). Multiple imputation was performed for missing values of change in score at each follow-up time prior to final data analysis. Twenty sets of imputed data for the changes outcome at each time were modeled using pre-treatment values of the outcome, age, gender, employment (yes/no), and treatment group as explanatory variables, using a chained equations approach.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Condition #1: PsychoEducation (ED) | Condition #2:Self-Hypnosis Training (HYP) | Condition #3: Mindfulness Meditation (MM)
Number analyzed (Participants) | 110 | 110 | 108
score on a scale | -.57 [-.63 to -.52] | -.61 [-.67 to -.56] | -.85 [-90 to -.79]
Statistical Analysis 1: Comparison: Condition #1: PsychoEducation (ED) vs Condition #2:Self-Hypnosis Training (HYP) vs Condition #3: Mindfulness Meditation (MM); Based on our prior work comparing similar interventions, assuming decreases in average pain intensity of 0.3 points (on a 0-10 scale) for ED, between 0.8 to 1.4 points for HYP, and between 0.6 to 1 for MM, with standard deviations (SD) ranging from 0.15 to 1, significance level of 0.05, and using ANOVA as the statistical method, we calculated that 80 participants per arm at immediate post-treatment would provide at least 80% power to detect between-groups differences as specified; Test type: Superiority; p = .39, ANOVA — Statistical significance was set at p=.05

2. Other Pre Specified Outcome: Change From Pre-Treatment in Average Pain Intensity on a 0-10 Numerical Rating Scale 3 Months Following End of Treatment
Description: An average of all of the 24-hour ratings (range=1-4 ratings) of average pain intensity was obtained over a period of one week during each assessment period, pre-treatment and 3 months following the end of treatment.
  Range: 0-10, 0='no pain' and 10 ='pain as bad as you can imagine'
  The difference between the two average scores from the different assessment periods (pre-treatment and 3 months following end of treatment) was computed by subtracting the pre-treatment score from the 3 months following end of treatment score, resulting in a change score. A negative value denotes a decrease in pain intensity between the two assessment periods, whereas a positive value denotes an increase.
Time Frame: Change in Average Pain Intensity from Pre-Treatment to 3 Months Following End of Treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Condition #1: PsychoEducation | Condition #2:Self-Hypnosis Training | Condition #3: Mindfulness Meditation
Number analyzed (Participants) | 110 | 110 | 108
score on a scale | -.48 [-.55 to -.42] | -.95 [-1.02 to -.88] | -.67 [-.74 to -.61]
Statistical Analysis 1: Comparison: Condition #1: PsychoEducation vs Condition #2:Self-Hypnosis Training vs Condition #3: Mindfulness Meditation; Test type: Superiority; p = .05, ANOVA — Statistical significance was set at p=.05

3. Other Pre Specified Outcome: Change From Pre-Treatment in Average Pain Intensity on a 0-10 Numerical Rating Scale 6 Months Following End of Treatment
Description: An average of all of the 24-hour ratings (range=1-4 ratings) of average pain intensity was obtained over a period of one week during each assessment period, pre-treatment and 6 months following the end of treatment.
  Range: 0-10, 0='no pain' and 10 ='pain as bad as you can imagine'
  The difference between the two average scores from the different assessment periods (pre-treatment and 6 months following end of treatment) was computed by subtracting the pre-treatment score from the 6 months following end of treatment score, resulting in a change score. A negative value denotes a decrease in pain intensity between the two assessment periods, whereas a positive value denotes an increase.
Time Frame: Change in Average Pain Intensity from Pre-Treatment to 6 Months Following End of Treatment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Condition #1: PsychoEducation | Condition #2:Self-Hypnosis Training | Condition #3: Mindfulness Meditation
Number analyzed (Participants) | 110 | 110 | 108
score on a scale | -.28 [-.34 to -.22] | -1.04 [-1.11 to -.98] | -.86 [-.92 to -.80]
Statistical Analysis 1: Comparison: Condition #1: PsychoEducation vs Condition #2:Self-Hypnosis Training vs Condition #3: Mindfulness Meditation; Test type: Superiority; p < .001, ANOVA — Statistical significance was set at p= .05

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each subject following enrollment until study completion, approximately 9-12 months.
Arm/Group | Condition #1: PsychoEducation | Condition #2:Self-Hypnosis Training | Condition #3: Mindfulness Meditation
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/110 | 0/108
Serious Adverse Events (participants affected / at risk) | 22/110 | 12/110 | 18/108
Other Adverse Events (participants affected / at risk) | 73/110 | 63/110 | 69/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Condition #1: PsychoEducation (N=110) | Condition #2:Self-Hypnosis Training (N=110) | Condition #3: Mindfulness Meditation (N=108)
New/Unusual/ Worsening Pain or Physical Discomfort At Least Possibly Related to Study Procedures (General disorders) | 1 (1) | 0 (0) | 0 (0)
Medically Important Surgery or Medical Procedure, Unrelated to Study Procedures (General disorders) | 13 (15) | 5 (5) | 6 (8)
New Cancer Diagnosis, Unrelated to Study Procedures (General disorders) | 1 (1) | 0 (0) | 0 (0)
Seizures, Unrelated to Study Procedures (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
New Physical Injury, Unrelated to Study Procedures (Injury, poisoning and procedural complications) | 2 (3) | 2 (2) | 3 (3)
Life Threatening Suicidal Ideation/Attempt, Unrelated to Study Procedures (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3)
Homicidal Ideation, Unrelated to Study Procedures (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Inpatient Hospitalization, Unrelated to Study Procedures (General disorders) | 1 (1) | 3 (3) | 3 (3)
Inpatient Hospitalization, Unrelated to Study Procedures (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Inpatient Hospitalization, Unrelated to Study Procedures (Cardiac disorders) | 1 (1) | 1 (2) | 1 (1)
Inpatient Hospitalization, Unrelated to Study Procedures (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inpatient Hospitalization, Unrelated to Study Procedures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Inpatient Hospitalization, Unrelated to Study Procedures (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Inpatient Hospitalization, Unrelated to Study Procedures (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Inpatient Hospitalization, Unrelated to Study Procedures (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
New/Unusual/ Worsening Pain or Physical Discomfort Unrelated to Study Procedures (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Condition #1: PsychoEducation (N=110) | Condition #2:Self-Hypnosis Training (N=110) | Condition #3: Mindfulness Meditation (N=108)
New Physical Injury, Unrelated to Study Procedures (General disorders) | 9 (10) | 13 (15) | 15 (20)
New/Unusual/ Worsening Nausea, At Least Possibly Related to EEG Procedures (General disorders) | 1 (1) | 0 (0) | 0 (0)
New/Unusual/ Worsening Nausea, At Least Possibly Related to Treatment Procedures (General disorders) | 0 (0) | 1 (1) | 0 (0)
New/Unusual/ Worsening Nausea, Unrelated to Study Procedures (General disorders) | 0 (0) | 0 (0) | 1 (1)
Adverse Medication Reaction, Unrelated to Study Procedures (General disorders) | 1 (1) | 2 (2) | 4 (4)
New Diagnosis, Not Life Threatening, Unrelated to Study Procedures (General disorders) | 0 (0) | 1 (1) | 1 (1)
New Illness/Infection/Untoward Medical Occurrence Unrelated to Study Procedures (General disorders) | 35 (60) | 31 (60) | 28 (41)
New Illness/Infection/Untoward Medical Occurrence, At Least Possibly Related to Treatment Procedures (General disorders) | 0 (0) | 2 (2) | 0 (0)
New/Unusual/ Worsening Cognitive Difficulties, Unrelated to Study Procedures (General disorders) | 0 (0) | 1 (1) | 1 (2)
New/Unusual/ Worsening Fatigue, Unrelated to Study Procedures (General disorders) | 3 (3) | 4 (5) | 4 (4)
New/Unusual/ Worsening Headache/Migraine, At Least Possibly Related to Study Self-Report Measures (General disorders) | 0 (0) | 0 (0) | 1 (1)
New/Unusual/ Worsening Headache/Migraine, At Least Possibly Related to EEG Procedures (General disorders) | 0 (0) | 1 (1) | 0 (0)
New/ Worsening Headache/Migraine, At Least Possibly Related to Baseline Hypnotizability Assessment (General disorders) | 0 (0) | 1 (1) | 0 (0)
New/Unusual/ Worsening Headache/Migraine, Unrelated to Study Procedures (General disorders) | 10 (11) | 10 (16) | 5 (7)
New/Unusual/ Worsening Pain or Physical Discomfort Unrelated to Study Procedures (General disorders) | 23 (36) | 21 (34) | 23 (42)
New/Worsening Psych. Discomfort At Least Possibly Related to Baseline Hypnotizability Assessment (General disorders) | 2 (2) | 4 (4) | 6 (6)
New/Worsening Psychological Discomfort At Least Possibly Related to Study Procedures, General (General disorders) | 1 (1) | 0 (0) | 0 (0)
New/Unusual/ Worsening Psychological Discomfort At Least Possibly Related to EEG Procedures (General disorders) | 2 (2) | 6 (6) | 3 (3)
New/Unusual/ Worsening Psychological Discomfort At Least Possibly Related to Self-Report Measures (General disorders) | 1 (1) | 3 (3) | 4 (5)
New/Unusual/ Worsening Psychological Discomfort At Least Possibly Related to Treatment Procedures (General disorders) | 1 (1) | 7 (8) | 3 (3)
New/Unusual/ Worsening Psychological Discomfort, Unrelated to Study Procedures (General disorders) | 7 (8) | 12 (16) | 11 (11)
New/Worsening Skin Irritation, At Least Possibly Related to Wearing Sleep Sub-Study Actigraph Device (General disorders) | 1 (1) | 5 (6) | 1 (1)
New/Unusual/ Worsening Sleep Problems, At Least Possibly Related to Sleep Sub-Study Procedures (General disorders) | 0 (0) | 0 (0) | 1 (1)
New/Unusual/ Worsening Sleep Problems, At Least Possibly Related to Treatment Procedures (General disorders) | 1 (1) | 0 (0) | 0 (0)
New/Unusual/ Worsening Sleep Problems Unrelated to Study Procedures (General disorders) | 2 (2) | 5 (5) | 3 (3)
New/Worsening Pain, Phys. Discomfort at Least Possibly Related to Baseline Hypno. Assessment (General disorders) | 7 (7) | 3 (3) | 2 (2)
New/Unusual/Worsening Pain or Physical Discomfort at Least Possibly Related to Consent Session (General disorders) | 0 (0) | 2 (2) | 0 (0)
New/Unusual/Worsening Pain or Physical Discomfort at Least Possibly Related to EEG Procedures (General disorders) | 8 (8) | 3 (3) | 4 (5)
New/Unusual/Worsening Pain or Physical Discomfort at Least Possibly Related to Self-Report Measures (General disorders) | 0 (0) | 0 (0) | 1 (1)
New/Unusual/Worsening Pain or Physical Discomfort at Least Possibly Related to Treatment Procedures (General disorders) | 1 (1) | 7 (7) | 8 (8)
Non-Life Threatening Suicidal Ideation, Unrelated to Study Procedures (General disorders) | 1 (1) | 0 (0) | 1 (1)
Non-Life Threatening/ Outpatient Surgery or Medical Procedure, Unrelated to Study Procedures (General disorders) | 22 (24) | 14 (20) | 18 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT02653664/Prot_SAP_002.pdf
  • Informed Consent Form (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT02653664/ICF_001.pdf